CLINICAL TRIAL: NCT02944916
Title: Pilot Study Evaluating the Use of a New Device for Transanal Irrigation in Patient With Bowel Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPM-G-H-1601; 2016-A00631-50 (Other: FRENCH HEALTH AUTORITY)
Record Dates: First submitted 2016-09-20; First posted 2016-10-26 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IryPump R Set (Experimental): A new set for transanal irrigation composed by 2 parts : 1 pump and 1 rectal catheter . 1 rectal catheter used per irrigation respecting the patient usual frequency of transanal irrigation
  Interventions: Device: IryPump R Set

INTERVENTIONS:
Device: IryPump R Set

SUMMARY:
The study descripted of efficacy of IryPump®R Set in term of success of the procedure at each irrigation

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old,
2. Patient having signed an informed consent
3. Patient having neurologic or non neurologic bowel disorders, being initiated to TAI and practicing TAI with Peristeen® for the management of her/his bowel disorders, for at least 6 weeks, with satisfying results.
4. Patient practicing TAI on the basis of 1 procedure/ week as a minimum or more frequently
5. Patient capable to perform the procedure of transanal irrigation himself or with the help of a caregiver
6. Patient having a mental capacity to participate to the study (i.e. to understand the study and to answer to the questions)
7. Patient agrees to test IryPump® Set R for a time corresponding to 5 consecutive irrigations and a maximum of 4 weeks.
8. Patient covered by social security

Exclusion Criteria:

1. Patient with bowel obstruction
2. Patient already participating in another clinical study or who have previously participated in this investigation,
3. Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Success of the trans anal irrigation (TAI) procedure | Duration of the study per patient will correspond to the realisation of 5 consecutive TAI in a maximum of 41 days of follow up
  The patient will practice TAI following his usual frequency (depending on his intestinal transit). After each TAI, the patient will evaluate the success of the procedure (defined as satisfying output evacuation of the bowel according to the patient usual pattern in term of volume of water instilled and absence of leakages between 2 irrigations).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Charvier, Principal Investigator — Henry Gabrielle Hospital- St Genis Laval- France